CLINICAL TRIAL: NCT04378530
Title: Mindfulness Takes Practice: mHealth Tools for Building Persistent Mindfulness Meditation Habits
Brief Title: Mindfulness Takes Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STUDY00011788
Record Dates: First submitted 2020-04-13; First posted 2020-05-07 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Stress; Habits
MeSH Terms: conditions — Habits

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Personalized Cue (Experimental): Participants in the intervention group will be recommended to participate in at least 10 minutes per day of meditation via a smartphone application for 8 weeks. Participants will receive anchoring specific push notifications and will respond to one, multiple-choice EMA (ecological momentary assessment) question 1x per day. Participants will be asked to select a cue to use to remember to meditate.
  Interventions: Behavioral: Personalized Anchoring Strategy
- Study control (Active Comparator): Participants in the control group will be recommended to participate in at least 10 minutes per day of meditation via a smartphone application for 8 weeks. Participants will receive non-anchoring specific push notifications and will respond to one, multiple-choice EMA (ecological momentary assessment) question 1x per day.
  Interventions: Behavioral: Non-Anchoring Strategy Control
- Fixed Cue (Experimental): Participants in the intervention group will be recommended to participate in at least 10 minutes per day of meditation via a smartphone application for 8 weeks. Participants will receive anchoring specific push notifications and will respond to one, multiple-choice EMA (ecological momentary assessment) question 1x per day. Participants will be given a specific cue (i.e. leaving the bathroom in the morning) to use to remember to meditate.
  Interventions: Behavioral: Fixed Anchoring Strategy

INTERVENTIONS:
Behavioral: Personalized Anchoring Strategy — The study will run for 8 weeks. Intervention participants will participate in the meditation features in their Calm account. Each participant will receive anchoring specific push notifications related to, tracking sessions completed, reminders, mood symptom tracking, and group-specific goal reminders. The intervention group will be provided an anchoring strategy video on the persistence of daily meditation practice and receive anchoring strategy specific push notification study reminders.
  Participants will be asked to choose a cue to use as an anchoring strategy. Health and well-being measures will be taken at baseline and post-intervention. Participation in the Calm meditations will be tracked (app feature used, time of day used, and time spent in meditation) by the Calm informatics team. Additionally, they will answer one, multiple choice EMA (ecological momentary assessment) question 1x per day (8am, 1pm or 6pm).
  Other Names: Personalized Cue
  Arms: Personalized Cue
Behavioral: Non-Anchoring Strategy Control — The study will run for 8 weeks. Control participants will participate in the meditation features in their Calm account. Each participant will receive non-anchoring specific push notifications related to, tracking sessions completed, reminders, mood symptom tracking, and group-specific goal reminders. The control group will not be provided an anchoring strategy video on the persistence of daily meditation practice and receive non-anchoring strategy specific push notification study reminders. Health and well-being measures will be taken at baseline and post-intervention. Participation in the Calm meditations will be tracked (app feature used, time of day used, and time spent in meditation) by the Calm informatics team. Additionally, they will answer one, multiple-choice EMA (ecological momentary assessment) question 1x per day (8am, 1pm or 6pm).
  Arms: Study control
Behavioral: Fixed Anchoring Strategy — The study will run for 8 weeks. Intervention participants will participate in the meditation features in their Calm account. Each participant will receive anchoring specific push notifications related to, tracking sessions completed, reminders, mood symptom tracking, and group-specific goal reminders. The intervention group will be provided an anchoring strategy video on the persistence of daily meditation practice and receive anchoring strategy specific push notification study reminders. Participants will be asked to use a cue given by the research team. Health and well-being measures will be taken at baseline and post-intervention. Participation in the Calm meditations will be tracked (app feature used, time of day used, and time spent in meditation) by the Calm informatics team. Additionally, they will answer one, multiple choice EMA (ecological momentary assessment) question 1x per day (8am, 1pm or 6pm).
  Other Names: Fixed Cue
  Arms: Fixed Cue

SUMMARY:
The purpose of the study is to optimize the delivery of mHealth tools to support the formation of persistent mindfulness meditation routines.

Aim 1: Identify the efficacy of the anchoring strategy on the persistence of daily meditation practice.

H1: Persistence (measured through repeated observations of panel regression models of the daily likelihood of mindfulness mediation over the 16-week follow-up period) will be greater among AG as compared to CG.

Aim 2: Determine participant phenotypes that are (a) associated with successfully anchoring daily meditation or (b) likely to need additional supports. Potential moderators of the anchoring strategy's success include participants' daily schedule, type of work, household composition, motivation, time and risk preferences, and prior exposure to mindfulness, which will be analyzed in the panel regression model framework above.

Aim 3: Determine the optimal type, timing, and sequence of push notifications for encouraging daily mindfulness meditation within and across study groups. The efficacy of each push notification type (tracking sessions completed, reminders, mood symptom tracking, and group-specific goal reminders), timing, and dynamics on the anchoring of daily meditation will inform a subsequent, just-in-time adaptive intervention (JITAI).

Impact: This study will inform an optimal JITAI R01 proposal that will personalize the type and temporal dynamics of app-based daily supports for successfully routinizing daily meditation, and determine its effects on mental health, specifically PTSD. Lifetime prevalence of PTSD is 7% in adults and meditation is known to reduce PTSD. If effective

DETAILED DESCRIPTION:
Recruitment: Participants will be recruited for a "health and well-being" study starting July, 2020. Interested participants will be directed to a Qualtrics link to complete an online eligibility screener. The screener will take approximately 3 minutes to complete (See Eligibility Survey). The survey will be free, voluntary, and available online. Participants will be allowed to skip questions in the survey.

Eligibility: Once eligibility is determined, eligible participants will be sent an informed consent. Ineligible participants will be sent an email notifying their status and why. Once an informed consent is signed and received, the participant will be notified of their random assignment and study start date. Participants will be randomized via an online randomizer (i.e., randomizer.com) to either the Anchor Group (intervention) or the control group.

Enrollment: The Research Team will email the participants instructions to download Calm (See Participant Scripts). On their study start date the participant will be sent their baseline questionnaires via a Qualtrics link. The measures will be online and should take approximately 20 minutes to complete (See Baseline Questionnaires).

Intervention: The study will run for 8-weeks. Intervention participants will receive access to the mobile application Calm and be recommended to participate in the meditation features. Each participant will receive push notifications related to, tracking sessions completed, reminders, mood symptom tracking, and group-specific goal reminders. The intervention group will be provided an anchoring strategy video on the persistence of daily meditation practice and receive anchoring strategy specific push notification study reminders. The control group will receive access to the mobile application Calm and be recommended to participate in the meditation features but will not be asked to watch the anchoring strategy video. The control group will also receive push notification reminders however, they will not be anchor strategy specific (See Push Notifications).

Tracking: Participation in the Calm meditations will be tracked (app feature used, time of day used, and time spent in meditation) by the Calm informatics team. Additionally, they will answer one, multiple-choice EMA (ecological momentary assessment) question each evening (see Study Questionnaires).

Post-study: Post-study questionnaires and the satisfaction survey will be emailed to intervention and control participants via a link from Qualtrics (See Post-study questionnaires). The post-intervention surveys will be online and take about 20 minutes and the satisfaction survey will take about 5 minutes.

Follow up: Participants will receive a follow up survey to complete via Qualtrics at 16 weeks. Follow up questionnaires and the satisfaction survey will be emailed to intervention and control participants via a link from Qualtrics. The follow up surveys will be online and take about 20 minutes and the satisfaction survey will take about 5 minutes. The follow up surveys will be identical to the post-study questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Men or Women
* Between 18 and 60 years of age
* Able to read/understand English
* Have access to a smartphone on a daily basis
* Reside in the US or a US territory
* Willing to be randomized
* Willing to download a mobile application
* Paid for Calm but do not use it OR paid for 60 days and then after 30 days no activity

Exclusion Criteria:

* Currently using the Calm app or another meditation app
* Currently participating in >60 mins of meditation/yoga in one month within the last 6 months.
* Currently reside outside the United States
* Email provided is not associated with Calm account

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 174 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Persistence of daily meditation | Change measured over study (8 weeks) and follow up (16 weeks) periods.
  Persistence of daily meditation will be measured using objective app usage data provided by the Calm app informatics. Data will be on daily meditation minutes and an indicator for any daily meditation. We will measure change in persistence in daily meditation throughout the study.

SECONDARY OUTCOMES:
Stress | Change from baseline (week 0) to post-intervention (week 8) to follow up (week 16)
  Stress will be measured using the Perceived Stress Scale -10 item, with scores ranging from 10-40) and a higher score indicates a worse outcome.
Anxiety | Change from baseline (week 0) to post-intervention (week 8) to follow up (week 16)
  Anxiety will be measured using the Hospital Anxiety and Depression Scale, with scores ranging from 0-21, and a higher score indicates a worse outcome.
Depression | Change from baseline (week 0) to post-intervention (week 8) to follow up (week 16)
  Depression will be measured using the Hospital Anxiety and Depression Scale, with scores ranging from 0-21, and a higher score indicates a worse outcome.
Global Health | Change from baseline (week 0) to post-intervention (week 8) to follow up (week 16)
  Global health will be measured using the PROMIS Global Health Scale v1.2, with scores ranging from 4-20, and higher scores indicate a better outcome.
PTSD | Change from baseline (week 0) to post-intervention (week 8) to follow up (week 16)
  PTSD will be measured using the Impact of Events Scale-Revised, with scores ranging from 0-88, with higher scores indicating a worse outcome.
Emotional Regulation | Change from baseline (week 0) to post-intervention (week 8) to follow up (week 16)
  Emotional regulation will be measured using the Difficulties in Emotional Regulation -18, with scores ranging from 18-90, with higher scores indicating a worse outcome.
HABIT | Change from baseline (week 0) to post-intervention (week 8) to follow up (week 16)
  Habit will be measured using the habit questionnaire scored is the sum across the four questions (which are individually scored from 1-5 based on degree of agreement), where a higher score indicates more behavioral automaticity (strong habit).
COVID-19 | Change from baseline (week 0) to post-intervention (week 8) to follow up (week 16)
  COVID-19 as a mediator to the other health and well-being measures will be measured through a COVID-19 questionnaire created by the researcher. The items are scored from 1-5 with higher scores indicating COVID as a more significant mediator.
Feasibility: Acceptability | Measured at post-intervention about experience in study (8 weeks) and follow up (16 weeks)
  Acceptability will be measured using a satisfaction survey at the end of the study, following all other measures (satisfied with the intervention and perceive daily meditation and app components as appropriate and useful)

CONTACTS AND LOCATIONS:
Overall Officials: Chad Stecher, PhD, Principal Investigator — Arizona State University
Locations (1):
- Arizona Biomedical Collaborative, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stecher C, Sullivan M, Huberty J. Using Personalized Anchors to Establish Routine Meditation Practice With a Mobile App: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2021 Dec 22;9(12):e32794. doi: 10.2196/32794. PMID 34941558